CLINICAL TRIAL: NCT06219226
Title: Hyperpure Chlorine Dioxide Versus Chlorhexidine in Intra-oral Halitosis (ODOR Trial)
Brief Title: Investigating the Effect of Chlorine Dioxide and Chlorhexidine Mouthwash on Bad Breath
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Eszter Á Szalai, DMD, Assistant lecturer, Semmelweis University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 838
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Halitosis
Keywords: ClO2; mouth rinse; malodor
MeSH Terms: conditions — Halitosis | interventions — chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chlorine dioxide mouthwash (Experimental): Participants will rinse once with hyper-pure ClO2 (0.003%) mouthwash.
  Interventions: Procedure: Chlorine dioxide mouthwash
- Chlorhexidine mouthwash (Active Comparator): Participants will rinse once with chlorhexidine-containing mouthwash (0.2%).
  Interventions: Procedure: Chlorhexidine mouthwash

INTERVENTIONS:
Procedure: Chlorine dioxide mouthwash — This one rinsing will last 2x15 seconds(2x12,5ml).
  Other Names: Solumium Coral®
  Arms: Chlorine dioxide mouthwash
Procedure: Chlorhexidine mouthwash — This one rinsing will last 2x15 seconds(2x12,5ml).
  Other Names: Curasept ADS 220, 0.2%
  Arms: Chlorhexidine mouthwash

SUMMARY:
The ODOR trial will be a single-centric, double-blinded, parallel-group, double-armed pilot randomized controlled trial with a non-inferiority design. The efficacy of hyperpure chlorine dioxide will be compared to chlorhexidine mouthwash. The short-term effect of the mouthwashes will be investigated in a 3-hour-long period. The primary endpoint will be the changes in the organoleptic testing scores.

DETAILED DESCRIPTION:
Eligible patients will be randomly allocated to two groups in a 1:1 ratio. Necessary data will be collected with prespecified electronic case report forms (REDCap). The statistician will calculate the sample size at the end of the pilot investigation of the first 30-30 patients. If feasible, investigators will continue the study by enrolling more patients.

ELIGIBILITY:
Inclusion Criteria:

* Organoleptic test score (OLS)>=2 for IOH
* Patients with at least 20 teeth
* 8 hours of scented oral hygiene product usage, 4 hours of eating, and 2 hours of drinking restriction
* on the day of investigation, restriction of alcohol, caffeine, perfume usage, and food intake with characteristic smell

Exclusion Criteria:

* Medical history of systematic and infectious diseases (e.g., hepatitis, HIV, tuberculosis).
* Antibiotic use within the month before the study's start or during the trial or any regular medication
* Extraoral halitosis (will be distinguished by observing the nasal breath)
* Eat foods (like garlic) linked to oral malodor on the day before and the sampling day, as well as wear heavily fragrant cosmetics on that day.
* Patients with removable dentures
* Smokers (Cigars, Cigarettes, Pipes, Chewing tobacco, e-cigarette, or vaping products used in the last month)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2025-12-18 (Estimated); Study Completion 2025-12-18 (Estimated)

PRIMARY OUTCOMES:
Changes of the organoleptic testing scores | immediately after the rinse and 3 hours later
  (gold standard 6-point (0-5) intensity scale. The examiner rates it 0 when the patient has no halitosis, and 5 when it is very severe)

SECONDARY OUTCOMES:
Changes of the volatile sulfur compounds | immediately after the rinse and 3 hours later
  with gas chromatography
Self-perceived halitosis | immediately after the rinse and 3 hours later
  with a visual analog scale ratings (0-100, 0 = No Pain, 100 = Worst Possible Pain)

OTHER OUTCOMES:
Side effects | immediately after the rinse and 3 hours later
  (e.g., tooth discoloration, signs of allergic reactions, subjective experiences: unpleasant taste, false taste or burning sensation, pain, changes in salivary flow)

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University, Budapest, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Szalai E, Tajti P, Szabo B, Hegyi P, Czumbel LM, Shojazadeh S, Varga G, Nemeth O, Keremi B. Daily use of chlorine dioxide effectively treats halitosis: A meta-analysis of randomised controlled trials. PLoS One. 2023 Jan 12;18(1):e0280377. doi: 10.1371/journal.pone.0280377. eCollection 2023. PMID 36634129
- [Background] Noszticzius Z, Wittmann M, Kaly-Kullai K, Beregvari Z, Kiss I, Rosivall L, Szegedi J. Chlorine dioxide is a size-selective antimicrobial agent. PLoS One. 2013 Nov 5;8(11):e79157. doi: 10.1371/journal.pone.0079157. eCollection 2013. PMID 24223899
- [Background] Kumbargere Nagraj S, Eachempati P, Uma E, Singh VP, Ismail NM, Varghese E. Interventions for managing halitosis. Cochrane Database Syst Rev. 2019 Dec 11;12(12):CD012213. doi: 10.1002/14651858.CD012213.pub2. PMID 31825092
- [Derived] Szalai EA, Teutsch B, Babay V, Galvacs A, Hegyi P, Harsfalvi P, Pal R, Varga G, Lohinai ZM, Keremi B. Hyperpure chlorine dioxide versus chlorhexidine in intra-oral halitosis (ODOR trial) - protocol of a double-blinded, double-arm, parallel non-inferiority pilot randomized controlled trial. BDJ Open. 2024 May 20;10(1):35. doi: 10.1038/s41405-024-00221-8. PMID 38769314